CLINICAL TRIAL: NCT00047411
Title: Home Automatic External Defibrillator Trial -- HAT
Brief Title: Home Use of Automatic External Defibrillators to Treat Sudden Cardiac Arrest
Acronym: HAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Philips Medical Systems (Industry); Laerdal Medical (Industry)
Responsible Party: Gust H. Bardy, MD, Seattle Institute for Cardiac Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 147; U01HL067972 (NIH)
Record Dates: First submitted 2002-10-03; First posted 2002-10-04 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-03

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Heart Diseases; Death, Sudden, Cardiac
Keywords: CPR, AED
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Heart Diseases; Death, Sudden, Cardiac | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intervention: Immediate notification of EMS by telephone and prompt initiation of CPR, in accordance with published Basic Life Support guidelines.
  Interventions: Other: Cardiopulmonary Resuscitation
- 2 (Experimental): Use of the AED first, in accordance with published guidelines for AED use, followed by a call to EMS and perform CPR as in the control group.
  Interventions: Device: Automatic External Defibrillation

INTERVENTIONS:
Other: Cardiopulmonary Resuscitation — Immediate notification of EMS by telephone and prompt initiation of CPR, in accordance with published Basic Life Support guidelines
  Arms: 1
Device: Automatic External Defibrillation — Use the AED first, in accordance with published guidelines for AED use, followed by a call to EMS and perform CPR as in the control group.
  Arms: 2

SUMMARY:
To compare home use of an automatic external defibrillator (AED) to the use of local emergency medical system in treating survivors of sudden cardiac arrest.

DETAILED DESCRIPTION:
BACKGROUND:

Sudden cardiac arrest (SCA) occurs every two minutes throughout the United States, with more than 70 percent occuring at home. Because survival falls 10 percent per minute over the first ten minutes, it is imperative to defibrillate as soon as possible. Public efforts cannot provide defibrillation fast enough in most cases. Physicians believe the initial shock is best done using readily available AEDs by family members who are only seconds from their loved one.

DESIGN NARRATIVE:

This study tests the central hypothesis that providing an AED for home use will improve survival beyond that achieved from the typical response to sudden cardiac arrest. An estimated 7,000 people who have had an anterior myocardial infarction will be randomly assigned to one of two groups: 1) a standard response to sudden cardiac arrest, entailing calling an emergency medical service (EMS) system and performing CPR, or 2) the addition of a home AED to the standard response. The standard response will be augmented and standardized by the provision of a video on how to respond to sudden cardiac arrest and how to perform CPR. The goal for the standard response will be immediate notification of EMS and prompt CPR. The goal for the AED group will be to shock the cardiac arrest victim up to three times immediately, if indicated by the AED, and call EMS and perform CPR as soon as possible and preferably within two minutes of collapse. Participants will be enrolled for more than two years and followed for an additional two years. The study will be performed at 200 cardiology clinics.

ELIGIBILITY:
Inclusion Criteria:

* History of anterior myocardial infarction
* Live-in spouse or companion willing to administer CPR or AED therapy plus CPR

Exclusion Criteria:

* Existing implantable cardiac defibrillator or AED
* Current candidate for an implantable cardiac defibrillator
* Current "Do Not Resuscitate" orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7001 (Estimated)
Dates: Start 2002-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
All-cause mortality (measured throughout the study) | Five interim analyses of the data were performed and reviewed by the DSMB

SECONDARY OUTCOMES:
Survival in the home from cardiac arrest and survival with AED use. | Five interim analyses of the data were performed and reviewed by the DSMB
Quality of life of the participants and their spouses (measured throughout the study) | Five interim analyses of the data were performed and reviewed by the DSMB

CONTACTS AND LOCATIONS:
Overall Officials: Gust H. Bardy, Study Chair — Seattle Institute for Cardiac Research
Locations (1):
- Seattle Institute for Cardiac Research, Seattle, Washington, United States

REFERENCES:
- [Derived] Mark DB, Anstrom KJ, McNulty SE, Flaker GC, Tonkin AM, Smith WM, Toff WD, Dorian P, Clapp-Channing NE, Anderson J, Johnson G, Schron EB, Poole JE, Lee KL, Bardy GH. Quality of life effects of automatic external defibrillators in the home: results from the Home Automatic External Defibrillator Trial (HAT). Am Heart J. 2010 Apr;159(4):627-634.e7. doi: 10.1016/j.ahj.2010.01.013. PMID 20362722
- [Derived] Bardy GH, Lee KL, Mark DB, Poole JE, Toff WD, Tonkin AM, Smith W, Dorian P, Packer DL, White RD, Longstreth WT Jr, Anderson J, Johnson G, Bischoff E, Yallop JJ, McNulty S, Ray LD, Clapp-Channing NE, Rosenberg Y, Schron EB; HAT Investigators. Home use of automated external defibrillators for sudden cardiac arrest. N Engl J Med. 2008 Apr 24;358(17):1793-804. doi: 10.1056/NEJMoa0801651. Epub 2008 Apr 1. PMID 18381485